CLINICAL TRIAL: NCT06362161
Title: Establishment of an Interdisciplinary Functional Neurological Disorder (FND) Treatment Program and Development of a Clinical Care Pathway for FND
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Aaron Fobian, Associate Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300011066
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Functional Neurological Disorder; Convulsion, Non-Epileptic; Functional Seizure
MeSH Terms: conditions — Conversion Disorder; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to help providers develop an interdisciplinary treatment pathway for functional neurological disorder (FND) at University of Alabama at Birmingham (UAB), and will involve psychiatry, speech therapy, physical therapy, and occupational therapy. The study will also help providers to evaluate the treatment pathway and publish results regarding the process and outcomes.

DETAILED DESCRIPTION:
Prospective Study: Adult patients, and pediatric patients and their parent/guardian who are referred to the UAB functional neurological disorder (FND) clinical pathway will be screened for eligibility. Overall 750 participants (250 adult patients, 250 pediatric patients and their parent/guardian) will be enrolled in the prospective study.

For patients for whom an FND inpatient consult has been requested, the consulting psychologist will screen eligible participants. For outpatient FND patients, the psychiatry FND clinic scheduling coordinator will screen patients for eligibility. Potential eligible participants will provide verbal consent during the screening phone call.

Once verbal consent has been obtained, participants will be given the pre-treatment survey questions (via email for outpatient referrals, via a tablet computer for inpatient consults). These surveys will be different for adult FND patients, children with FND, and parents/guardians of children with FND; each survey will contain the appropriate consent/assent form. Participants will complete the pre-treatment surveys once they sign the appropriate consent/assent form.

During each outpatient visit with a clinician, patients will be administered the one-item Clinical Global Improvement Scale and asked about retrospective symptom frequency, which will be entered directly into the electronic health record (EHR). If patients are seeing physical, occupational, or speech therapy (PT/OT/Speech), the clinician will enter clinical measures directly into the EHR. Following the course of FND treatment, participants and parents/guardians (where applicable) will complete the post-survey questionnaires.

Participants may be asked to provide full facial pictures and/or videos before treatment and after treatment.

Retrospective study: EHR data of participants who recieved FND treatment at UAB FND clinical pathway from Jan 2020 to May 2023 will be collected retrospectively. 500 records will be screened for potential inclusion in the study. Overall, data will be extracted from 350 patient records.

The research team will utilize EHR entries to pull any clinical data related to FND treatment visits (inpatient consults, outpatient psychiatry/PT/OT/Speech). This EHR data collection will be both retrospective and prospective, and include all records related to FND treatment, including neurology, PT/OT/Speech, and psychiatry notes.

The cost of participant's standard medical care will be billed to them and/or their insurance company in the usual manner. Participants will not be paid for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FND
* Can read and write English fluently
* Referred to UAB outpatient treatment for FND in physical, occupational, or speech therapy
* Referred to UAB outpatient treatment for FND in psychiatry
* Referred to inpatient consult for FND at Children's of Alabama or UAB Hospital
* Parent/guardian willing to participate in the study with a pediatric patient

Exclusion Criteria:

* Unable to read or write English fluently

Ages: 8 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be referred to the interdisciplinary FND clinical pathway via UAB- or non-UAB clinicians and physicians. Individuals who are referred will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Demographic Information | 4 months
  Includes questions regarding patient's demographic information, referring physician, current symptoms, medical history, and recent functioning including work and school missed, mobility aids used, or receipt of disability service. Completed by adult FND patients and parent/guardian of pediatric FND patients during the intake therapy session before beginning treatment and after completing FND treatment.
Hospital Anxiety and Depression Scale (HADS) | 4 months
  HADS is a self-assessment scale for detecting states of depression and anxiety in the setting of an outpatient hospital. Score ranges from 0-21 for depression and anxiety respectively and higher scores indicate greater anxiety and depression. Completed by adult patient before beginning treatment and after completing treatment.
ASM 121 functional assessment definitions | 4 months
  Assesses activities of daily living. Scores ranges from 12-60; higher scores indicate greater difficulty in performing daily activities. Completed by adult patient before beginning treatment and after completing treatment.
SF-36 (subjective health and wellbeing) | 4 months
  Assesses physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Completed by adult patient before beginning treatment and after completing treatment.
Work and Social Adjustment Scale (WSAS) | 4 months
  Assesses impairment in functioning. Score ranges from 0-40; higher scores indicate severe functional impairment. Completed by adult patient before beginning treatment and after completing treatment.
Patient Health Questionnaire 15 | 4 months
  Assesses patient's physical symptom severity. Scores ranges from 0-30; higher scores indicate severe somatoform disorder. Completed by adult patient before beginning treatment and after completing treatment.
Dizziness Handicap Inventory | 4 months
  Assesses functional, physical and emotional problems related to dizziness, specifically considering their condition in the last month. Scores range from 0-100; higher scores indicate severe handicap. Completed by adult FND patient and pediatric patients and their parent/guardian before beginning treatment and after completing treatment.
Dizziness Symptom Profile | 4 months
  Assesses severity of dizziness. Score ranges from 0-124; higher scores indicate severe impairment due to dizziness. Completed by adult patient, and pediatric patient and their parent/guardian before beginning treatment and after completing treatment.
Adult Tic Questionnaire (ATQ) | 4 months
  The ATQ is a brief self-report questionnaire that provides information regarding frequency, intensity, and severity of vocal and motor tics. Completed by adult patient before beginning treatment and after completing treatment.
Child Self-Report Tic Questionnaire | 4 months
  The child self-report tic questionnaire is a brief self-report questionnaire that provides information regarding frequency, intensity, and severity of vocal and motor tics.Completed by pediatric patient before beginning treatment and after completing treatment.
Parent Tic Questionnaire (PTQ) | 4 months
  The PTQ assesses tic severity, frequency and intensity in the past week, allowing for individual parent ratings of tic presence or absence for 14 vocal tics and 14 motor tics.Completed by parent/guardian of pediatric patients before beginning treatment and after completing treatment.
Seizure Questionnaire | 4 months
  Assesses any functional seizure the patient is experiencing. Completed by adult FND patients, pediatric patients and their parent/guardian before beginning treatment and after completing FND treatment.
Level 2-Somatic Symptom report | 4 months
  Measures symptom severity in children; scores ranges from 0-26, higher scores indicate greater symptom severity. Completed by pediatric patient and parent/guardian before beginning treatment and after completing treatment.
Revised Children's Anxiety and Depression Scale (RCADS) | 4 months
  Measures anxiety and depression symptoms in children; total score ranges from 0-141, higher scores indicate increased symptom severity. Completed by pediatric patient and parent/guardian before beginning treatment and after completing treatment.
Functional Disability Inventory (FDI) | 4 months
  Measures physical functioning and disability in children with chronic pain; score ranges from 0-60, higher scores indicate greater perceived functional disability. Completed by pediatric patient and parent/guardian before beginning treatment and after completing treatment.
Impact on the Family Scale | 4 months
  Assesses parental perceptions of the impact of a child's medical condition on the family (assesses impact on financial burden, familial/social impact, personal strain and mastery); higher scores indicate greater financial burden on the family. Completed by pediatric patient and parent/guardian before beginning treatment and after completing treatment.
Pediatric Quality of Life (Peds-QL) | 4 months
  Assesses quality of life, greater scores indicate greater quality of life. Scores range from 0-100. Completed by pediatric patient and parent/guardian before beginning treatment and after completing treatment.
Healthcare Utility Questionnaire | 4 months
  Assesses patients visits to a physician's office or emergency room related to their FND symptoms. Completed by adult patient, and pediatric patient and their parent/guardian throughout the study.
Assessment of control over symptoms | 4 months
  Single question that assesses the control patients have over their symptoms. Completed by adult patient, and pediatric patient and their parent/guardian before beginning treatment and after completing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fobian, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States